CLINICAL TRIAL: NCT05682144
Title: A Phase I Open Label Study to Evaluate the Safety and Tolerability of ISP-001 in Adult Patients With Mucopolysaccharidosis Type I Hurler-Scheie and Scheie
Brief Title: ISP-001: Sleeping Beauty Transposon-Engineered B Cells for MPS I
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Immusoft of CA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT2021-24
Record Dates: First submitted 2022-12-12; First posted 2023-01-12 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Mucopolysaccharidosis IH/S; Mucopolysaccharidosis IS
Keywords: MPS IH/S; MPS IS
MeSH Terms: conditions — Mucopolysaccharidosis I

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Autologous Plasmablasts (B cells) (Experimental): Dose Level: 5 x 10e7 cells/kg on Day 0
  Interventions: Biological: Autologous Plasmablasts (B cells)

INTERVENTIONS:
Biological: Autologous Plasmablasts (B cells) — Autologous plasmablasts (B cells) engineered to express α-L-iduronidase (IDUA) using the Sleeping Beauty (SB) transposon system.

SUMMARY:
A first-in-human study using ISP-001 in adult patients with Mucopolysaccharidosis Type I Hurler-Scheie and Scheie.

DETAILED DESCRIPTION:
This is a Phase 1, first-in-human, open-label, single-arm study in which adult patients with Mucopolysaccharidosis Type I Hurler-Scheie and Scheie are treated with autologous plasmablasts engineered to express α-L-iduronidase (IDUA) using the Sleeping Beauty transposon system (ISP-001). This study will evaluate the safety and tolerability of ISP-001.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Mucopolysaccharidosis type I Hurler-Scheie or Scheie syndrome.
* Age ≥ 18 years at time of study registration.
* Creatinine clearance, calculated or measured directly, that is >60ml/min/1.73m2.
* Ejection fraction ≥ 40% by echocardiogram.
* Must commit to traveling to the study site for the necessary follow-up evaluations.
* Must agree to stay <45-minute drive from the study site for a minimum of 5 days after cell infusion.

Exclusion Criteria:

* Known familial inherited cancer syndrome. Suspected cases will be investigated, per the physicians discretion, using relevant genetic tests to determine presence of germline mutations.
* History of B cell related cancer, EBV lymphoproliferative disease or autoimmune disorders.
* Evidence of active graft-vs-host disease.
* Underwent a previous hematopoietic stem cell transplant (HSCT).
* Requirement for systemic immune suppression.
* Requirement for continuous supplemental oxygen.
* Any medical condition likely to interfere with assessment of safety or efficacy of the study treatment.
* In the investigator's judgement, the subject is unlikely to complete all protocol-required study visits or procedures, including follow up visits, or comply with the study requirements for participation.

Other protocol defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2039-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events and serious adverse events | 24 Weeks
  Incidence of Adverse Events as assessed by CTCAE (v 5.0)

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events and serious adverse events | 48 Weeks
  Incidence of Adverse Events as assessed by CTCAE (v 5.0)
Determination of Absolute Numbers of B and T cell populations | 1Year
  Determination of Absolute Numbers of B and T cell populations in peripheral blood at baseline and at scheduled time points post infusion.
Concentration of IDUA | 1 Year
  Determine IDUA concentration in plasma at baseline and at scheduled time points post infusion.
Assessment of Storage Material (glycosaminoglycan, or GAG) | 1 Year
  Assessment of Storage Material (glycosaminoglycan, or GAG) in urine at baseline and at scheduled time points post infusion.
Levels of Circulating Antibodies (IgG, IgM, IgA, and IgE) | 1 Year
  Determine levels of circulating antibodies (IgG, IgM, IgA, and IgE) at baseline and at scheduled time points post infusion.
Analysis of PBMCs | 1 Year
  PBMCs will be analyzed at baseline and at scheduled time points post infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Immusoft Clinical Development, Study Director — Immusoft of CA, Inc.
Locations (2):
- United States (2):
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - University of Minnesota, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No